CLINICAL TRIAL: NCT04221698
Title: Do Young Triathletes Have a Greater Predisposition to Suffer Running Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J.J. Amer-Cuenca (Other)
Responsible Party: Sponsor-Investigator, J.J. Amer-Cuenca, Vice Dean, Cardenal Herrera University
Organization: Cardenal Herrera University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CEI18/137
Record Dates: First submitted 2019-12-19; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Gait Retraining; Kinematics
Keywords: Gait Analysis; Triathlon; Running; Gait Retraining

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait Retraining Group (Experimental): Athletes from the Triathlon Plan in High Performance of the Valencian Community in Spain performing individual gait retraining sessions
  Interventions: Other: Gait retraining

INTERVENTIONS:
Other: Gait retraining — 5 gait retraining sessions of continuous feedback in real time during running sessions; using videotape feedback, a digital metronome to increase step rate, and verbal feedback to reduce the tendency to heel strike upon ground contact. Verbal feedback is offered during the 25- to 30-minute running sessions following a series of drills aimed at improving running mechanics.

SUMMARY:
In running 70% of the lower limb, injuries are produced in the running segment. The vast majority of sports-related musculoskeletal injuries in young athletes are caused by overuse. Previous research has shown a clear association between running-related injuries and kinematic patterns, showing the existence of a causal relationship between biomechanical alterations and injures.

According to the evidence, that real-time visual and auditory feedback based on gait retraining should be considered to treat injured runners or prevent injuries. However, no previous studies have been carried out on whether gait retraining decreases running-related injuries incidence in young triathletes.

The investigators propose a study to determine the effect of gait retraining on the decrease in the number of running-related injuries and improve the running efficiency in young triathletes.

ELIGIBILITY:
Inclusion Criteria:

* Triathletes included in the Triathlon Plan in High Performance of the Valencian Community in Spain.
* Reported running a minimum of 2 days per week for the last 3 months with no reported injury.
* Worst pain rated a minimum of 3 out 10 on a numerical rating scale (NRS) for pain (0=no pain, 10=worst possible pain)

Exclusion Criteria:

* Previous musculoskeletal surgery.
* Neurological impairment
* Structural deformity in the knee.
* Pain suffered by trauma or sports activity, having stopped running or receiving additional treatment outside the study.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Surface Electromyography | Baseline - 7 months
  Mean activation amplitude of gluteus medius.

SECONDARY OUTCOMES:
3D Kinematic Analysis | Baseline - 7 months
  Peak angle at midstance defined as of the maximum pelvis joint angle between initial contact and toe-off. The tool to assess this variable would be an Inertial measurement unit (IMU) located at sacral vertebra S1
Maximal Oxygen Consumption (VO2max) | Baseline - 7 months
  Oxygen Consumption during running

OTHER OUTCOMES:
Self-report Questionnaire about Running-related injuries | Baseline - 7 months
  By means of a self-report questionnaire according to previous research in triathletes to document the incidence of overuse injuries previous and post gait retraining protocol season. Higher scores (number of injuries) mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martínez-Gramage, PhD, Principal Investigator — CEU Cardenal Herrera University
Locations (1):
- Juan J. Amer-Cuenca, Alfara del Patriarca, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bramah C, Preece SJ, Gill N, Herrington L. A 10% Increase in Step Rate Improves Running Kinematics and Clinical Outcomes in Runners With Patellofemoral Pain at 4 Weeks and 3 Months. Am J Sports Med. 2019 Dec;47(14):3406-3413. doi: 10.1177/0363546519879693. Epub 2019 Oct 28. PMID 31657964
- [Result] Bramah C, Preece SJ, Gill N, Herrington L. Is There a Pathological Gait Associated With Common Soft Tissue Running Injuries? Am J Sports Med. 2018 Oct;46(12):3023-3031. doi: 10.1177/0363546518793657. Epub 2018 Sep 7. PMID 30193080